CLINICAL TRIAL: NCT02431364
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Sequential, Dose-Escalating Trial to Evaluate the Safety and Tolerability of Oral Verdinexor (KPT-335) in Healthy Adult Subjects
Brief Title: Trial of Safety and Tolerability of Oral Verdinexor (KPT-335) in Healthy Adults
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administrative reason
Sponsor: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: KCP-335-701
Record Dates: First submitted 2015-04-22; First posted 2015-05-01 (Estimated); Results first posted 2021-04-13 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Healthy
Keywords: KPT-335; Verdinexor; Karyopharm; First-in-Human; Adult Subjects
MeSH Terms: interventions — verdinexor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Participants received matched placebo tablets to verdinexor tablets orally once daily on Days 1 and 3.
  Interventions: Other: Placebo
- Verdinexor 5 mg (Experimental): Participants received verdinexor 5 milligrams (mg) (2 tablets of 2.5 mg each) orally once daily on Days 1 and 3.
  Interventions: Drug: Verdinexor
- Verdinexor 10 mg (Experimental): Participants received verdinexor 10 mg tablet orally once daily on Days 1 and 3.
  Interventions: Drug: Verdinexor
- Verdinexor 20 mg (Experimental): Participants received verdinexor 20 mg tablet (2 tablets of 10 mg each) orally once daily on Days 1 and 3.
  Interventions: Drug: Verdinexor
- Verdinexor 40 mg (Experimental): Participants received verdinexor 40 mg tablet (4 tablets of 10 mg each) orally once daily on Days 1 and 3.
  Interventions: Drug: Verdinexor

INTERVENTIONS:
Drug: Verdinexor — Participants received verdinexor; Dosage form: coated, immediate release Tablet; Route of administration: oral
  Other Names: KPT-335
  Arms: Verdinexor 10 mg; Verdinexor 20 mg; Verdinexor 40 mg; Verdinexor 5 mg
Other: Placebo — Participants received placebo matched to verdinexor; Dosage form: coated, immediate release Tablet; Route of administration: oral
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, sequential, dose-escalation, Phase 1 trial to evaluate the safety and tolerability of verdinexor. Verdinexor or placebo will be given on Days 1 and 3 to healthy adult participants.

DETAILED DESCRIPTION:
This is a randomized, double-blind, sequential, dose-escalation, Phase 1 trial to evaluate the safety and tolerability of verdinexor. Verdinexor or placebo will be given on Days 1 and 3 to healthy adult participants.

Cohorts of 8 participants each (6 active, 2 placebo) will be sequentially administered verdinexor or placebo (one dose on Day 1 and one dose on Day 3) using a dose-escalation scheme. A conservative, sequential, dose-escalation strategy employing decreasing escalation increments will be used.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be in good health as determined by the investigator, based on the medical history, ECG, physical examination, and safety laboratory tests at screening.
* Participants must be identified as a non-smoker at the screening visit (a non-smoker is defined as an individual who has abstained from smoking for at least 1 year prior to the screening visit and who has a ≤ 15 pack year history of lifetime cigarette use). A urine cotinine test will be performed at screening and at the time of clinic check-in prior to study drug treatment.

Exclusion Criteria:

* The participant has any surgical or medical condition that potentially may alter the absorption, metabolism, or excretion of the study drug such as gastrectomy, Crohn's disease, or liver disease.
* The participant has a history of clinically significant allergies. Hay fever is allowed unless it is active or has required treatment within the previous 2 months.
* Presence of a chronic condition(s) with clinical or historical evidence of recent exacerbation, or other information to suggest non-control of such condition(s).
* History of alcohol abuse or drug addiction within 12 months of the screening visit.
* Any participant with active cataracts or medical history of cataracts.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2015-05-26 (Actual); Primary Completion 2015-10-01 (Actual); Study Completion 2015-10-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at single site in Australia from 26 May 2015 to 1 October 2015.
Pre-assignment Details: A total of 33 participants were enrolled and randomized, of which 1 participant randomized to verdinexor 20 milligrams (mg) arm discontinued the study before the start of the treatment (due to Adverse event [AE] prior to the pre-dose assessment). Total 32 participants started the study treatment.
Period: Overall Study
Arm/Group | Placebo | Verdinexor 5 mg | Verdinexor 10 mg | Verdinexor 20 mg | Verdinexor 40 mg
Started | 8 | 6 | 6 | 7 | 6
Treated | 8 | 6 | 6 | 6 | 6
Completed | 8 | 5 | 6 | 6 | 6
Not Completed | 0 | 1 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0
Not completed — Randomized but never treated | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who received at least one dose of verdinexor or placebo.
Groups:
- Verdinexor 5 mg: Participants received verdinexor 5 mg (2 tablets of 2.5 mg each) orally once daily on Days 1 and 3.
- Total: Total of all reporting groups
Arm/Group | Placebo | Verdinexor 5 mg | Verdinexor 10 mg | Verdinexor 20 mg | Verdinexor 40 mg | Total
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.0 (3.93) | 24.0 (3.35) | 26.5 (1.64) | 26.3 (6.09) | 27.8 (4.07) | 26.4 (4.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 4 | 5 | 5 | 22
  Male | 3 | 3 | 2 | 1 | 1 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 8 | 4 | 6 | 6 | 6 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 7 | 5 | 5 | 3 | 6 | 26
  Race: Asian | 0 | 0 | 1 | 2 | 0 | 3
  Race: Other | 1 | 1 | 0 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An AE was defined as the appearance of (or worsening of any pre-existing) undesirable sign, symptom, or medical condition that occur after participant's signed informed consent obtained. A serious adverse event (SAE) was defined as any AE, occurring at any dose (including after the informed consent form was signed and prior to dosing) that and regardless of causality that: results in death, was life-threatening (participant was at immediate risk of death from event as it occurred), requires in-patient hospitalization (formal admission to a hospital for medical reasons) or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect. TEAE was defined as any AE with onset or worsening of a pre-existing condition on or after the first administration of study treatment through 30 days following last dose or any event considered drug-related by the investigator through the end of the study.
Time Frame: From start of study drug administration up to Day 33
Population: Safety population included all participants who received at least 1 dose of verdinexor or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Verdinexor 5 mg | Verdinexor 10 mg | Verdinexor 20 mg | Verdinexor 40 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
Participants
  Participants with TEAEs | 5 | 6 | 3 | 4 | 5
  Participants with TESAEs | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to the Last Non-zero Concentration (AUC0-t) of Verdinexor
Description: AUC0-t was defined as area under the concentration-time curve from time zero to the last non-zero concentration
Time Frame: Days 1 and 3: pre-dose, 15 minutes, 30 minutes, 1, 2, 3, 4, 8, 12, 24, 48 (only for Day 3) hours post-dose
Population: Pharmacokinetic (PK) population included all participants who received at least 1 dose of verdinexor, had a pre-dose (baseline) blood draw, and had at least 1 qualified (above the limit of quantification [LOQ]) post-dose PK sample. Here, 'number analyzed' signifies number of participants evaluable at specific time points.
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Verdinexor 5 mg | Verdinexor 10 mg | Verdinexor 20 mg | Verdinexor 40 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
nanogram*hour per milliliter (ng*h/mL)
  Day 1 | 215 (34.2) | 445 (69.9) | 862 (129.6) | 1,856 (343.9)
  Day 3: number analyzed (Participants) | 5 | 6 | 6 | 6
  Day 3 | 196 (34.3) | 440 (103.4) | 991 (218.1) | 2,072 (521.6)

3. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Extrapolated to Infinity (AUC0-inf) of Verdinexor
Description: AUC0-inf was defined as area under the concentration-time curve from time zero to infinity (extrapolated). It was calculated as AUC0-t + Ct/kel, where: Ct = the last observed non-zero concentration, kel = elimination rate constant.
Time Frame: Days 1 and 3: pre-dose, 15 minutes, 30 minutes, 1, 2, 3, 4, 8, 12, 24, 48 (only for Day 3) hours post-dose
Population: PK population included all participants who received at least 1 dose of verdinexor, had a pre-dose (baseline) blood draw, and had at least 1 qualified (above the LOQ post-dose PK sample. Here, 'number analyzed' signifies number of participants evaluable at specific time points.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Verdinexor 5 mg | Verdinexor 10 mg | Verdinexor 20 mg | Verdinexor 40 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng*h/mL
  Day 1 | 235 (34.3) | 499 (75.1) | 991 (145.0) | 2,137 (371.0)
  Day 3: number analyzed (Participants) | 5 | 6 | 6 | 6
  Day 3 | 218 (31.6) | 491 (104.8) | 1,052 (217.6) | 2,141 (539.4)

4. Secondary Outcome: Maximum Observed Concentration (Cmax) of Verdinexor
Description: Cmax was defined as maximum observed concentration, taken directly from the plasma concentration data.
Time Frame: Days 1 and 3: pre-dose, 15 minutes, 30 minutes, 1, 2, 3, 4, 8, 12, 24, 48 (only for Day 3) hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Verdinexor 5 mg | Verdinexor 10 mg | Verdinexor 20 mg | Verdinexor 40 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
nanogram per milliliter (ng/mL)
  Day 1 | 27.8 (7.48) | 65.0 (12.13) | 122 (26.3) | 212 (81.6)
  Day 3: number analyzed (Participants) | 5 | 6 | 6 | 6
  Day 3 | 24.8 (5.42) | 56.2 (12.94) | 116 (36.9) | 252 (74.6)

5. Secondary Outcome: Average Plasma Concentration From Time Zero to 24 Hours Post-dose (Cavg0-24h) of Verdinexor
Description: Cavg0-24h was defined as average plasma concentration from time zero to 24 hours post-dose.
Time Frame: Days 1 and 3: pre-dose, 15 minutes, 30 minutes, 1, 2, 3, 4, 8, 12, 24 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Verdinexor 5 mg | Verdinexor 10 mg | Verdinexor 20 mg | Verdinexor 40 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng/mL
  Day 1 | 8.35 (1.835) | 19.6 (2.71) | 42.3 (9.97) | 72.4 (25.63)
  Day 3: number analyzed (Participants) | 5 | 6 | 6 | 6
  Day 3 | 8.73 (3.281) | 17.3 (4.91) | 44.4 (9.05) | 86.7 (29.56)

6. Secondary Outcome: Time of First Observation of Maximum Observed Concentration (Tmax) of Verdinexor
Description: Tmax was defined as time of first observation of Cmax, taken directly from the plasma concentration data.
Time Frame: Days 1 and 3: pre-dose, 15 minutes, 30 minutes, 1, 2, 3, 4, 8, 12, 24, 48 (only for Day 3) hours post-dose
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | Verdinexor 5 mg | Verdinexor 10 mg | Verdinexor 20 mg | Verdinexor 40 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
hours
  Day 1 | 3.0 [2.0 to 4.0] | 4.0 [2.0 to 4.0] | 3.0 [2.0 to 4.0] | 4.0 [2.0 to 4.0]
  Day 3: number analyzed (Participants) | 5 | 6 | 6 | 6
  Day 3 | 3.0 [2.0 to 4.0] | 3.0 [3.0 to 4.0] | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 4.0]

7. Secondary Outcome: Elimination Rate Constant (Kel) of Verdinexor
Description: Elimination rate constant was calculated using linear regression on the terminal portion of the log-linear concentration versus time curve.
Time Frame: Days 1 and 3: pre-dose, 15 minutes, 30 minutes, 1, 2, 3, 4, 8, 12, 24, 48 (only for Day 3) hours post-dose
Population: PK population included all participants who received at least 1 dose of verdinexor, had a pre-dose (baseline) blood draw, and had at least 1 qualified (above the LOQ) post-dose PK sample. Here, 'number analyzed' signifies number of participants evaluable at specific time points.
Measure: Mean (Standard Deviation); unit: per hour (1/h)
Arm/Group | Verdinexor 5 mg | Verdinexor 10 mg | Verdinexor 20 mg | Verdinexor 40 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
per hour (1/h)
  Day 1 | 0.113 (0.0314) | 0.091 (0.0227) | 0.082 (0.0177) | 0.097 (0.0306)
  Day 3: number analyzed (Participants) | 5 | 6 | 6 | 6
  Day 3 | 0.103 (0.0282) | 0.087 (0.0218) | 0.090 (0.0381) | 0.093 (0.0215)

8. Secondary Outcome: Elimination Half-life (t1/2) of Verdinexor
Description: t1/2 was defined as elimination half-life, it was calculated as ln(2)/kel.
Time Frame: Days 1 and 3: pre-dose, 15 minutes, 30 minutes, 1, 2, 3, 4, 8, 12, 24, 48 (only for Day 3) hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Verdinexor 5 mg | Verdinexor 10 mg | Verdinexor 20 mg | Verdinexor 40 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
hours
  Day 1 | 6.6 (1.97) | 8.0 (1.99) | 9.0 (2.68) | 7.8 (2.54)
  Day 3: number analyzed (Participants) | 5 | 6 | 6 | 6
  Day 3 | 7.3 (2.85) | 8.3 (1.91) | 8.7 (2.97) | 7.7 (1.76)

9. Secondary Outcome: Apparent Total Body Clearance (Cl/F) of Verdinexor
Description: Apparent total body clearance was calculated as Dose/AUC0-inf, uncorrected for fraction absorbed; reported normalized by participant body weight (kilogram [kg]).
Time Frame: Days 1 and 3: pre-dose, 15 minutes, 30 minutes, 1, 2, 3, 4, 8, 12, 24, 48 (only for Day 3) hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: liter per hour per kilogram (L/h/kg)
Arm/Group | Verdinexor 5 mg | Verdinexor 10 mg | Verdinexor 20 mg | Verdinexor 40 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
liter per hour per kilogram (L/h/kg)
  Day 1 | 0.32 (0.075) | 0.30 (0.023) | 0.31 (0.057) | 0.32 (0.040)
  Day 3: number analyzed (Participants) | 5 | 6 | 6 | 6
  Day 3 | 0.35 (0.068) | 0.30 (0.039) | 0.30 (0.059) | 0.33 (0.102)

10. Secondary Outcome: Apparent Volume of Distribution (Vd/F) of Verdinexor
Description: Vd/F was calculated as Dose/ (kel *AUC0-inf), uncorrected for fraction absorbed; reported normalized by participant body weight (kg).
Time Frame: Days 1 and 3: pre-dose, 15 minutes, 30 minutes, 1, 2, 3, 4, 8, 12, 24, 48 (only for Day 3) hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: liter per kilogram (L/kg)
Arm/Group | Verdinexor 5 mg | Verdinexor 10 mg | Verdinexor 20 mg | Verdinexor 40 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
liter per kilogram (L/kg)
  Day 1 | 3.0 (0.96) | 3.4 (0.89) | 3.9 (0.52) | 3.5 (1.01)
  Day 3: number analyzed (Participants) | 5 | 6 | 6 | 6
  Day 3 | 3.6 (1.13) | 3.6 (0.46) | 3.6 (0.90) | 3.7 (1.72)

11. Secondary Outcome: Accumulation Factor (AR) of Cmax
Description: An AR was defined as a ratio of mean of Cmax Day 3/ Cmax Day 1 for plasma verdinexor.
Time Frame: Days 1 and 3: pre-dose, 15 minutes, 30 minutes, 1, 2, 3, 4, 8, 12, 24, 48 (only for Day 3) hours post-dose
Population: PK population included all participants who received at least 1 dose of verdinexor, had a pre-dose (baseline) blood draw, and had at least 1 qualified (above the LOQ post-dose PK sample. Here 'number analyzed' signifies number of participants evaluable at specific time points.
Measure: Number; unit: Ratio
Arm/Group | Verdinexor 5 mg | Verdinexor 10 mg | Verdinexor 20 mg | Verdinexor 40 mg
Number analyzed (Participants) | 5 | 6 | 6 | 6
Ratio | 0.9 | 0.9 | 0.9 | 1.2

12. Secondary Outcome: Accumulation Factor (AR) of Cavg0-24Hour
Description: An AR was defined as a ratio of mean of Cavg0-24hour Day 3/ Cavg0-24hour Day 1 for plasma verdinexor.
Time Frame: Days 1 and 3: pre-dose, 15 minutes, 30 minutes, 1, 2, 3, 4, 8, 12, 24 hours post-dose
Population: as for outcome 11
Measure: Number; unit: Ratio
Arm/Group | Verdinexor 5 mg | Verdinexor 10 mg | Verdinexor 20 mg | Verdinexor 40 mg
Number analyzed (Participants) | 5 | 6 | 6 | 6
Ratio | 1.0 | 0.9 | 1.1 | 1.2

13. Secondary Outcome: Accumulation Factor (AR) of AUC0-t
Description: An AR factor was defined as a ratio of mean of AUC0-t Day 3/ AUC0-t Day 1 for plasma verdinexor.
Time Frame: Days 1 and 3: pre-dose, 15 minutes, 30 minutes, 1, 2, 3, 4, 8, 12, 24, 48 (only for Day 3) hours post-dose
Population: as for outcome 11
Measure: Number; unit: Ratio
Arm/Group | Verdinexor 5 mg | Verdinexor 10 mg | Verdinexor 20 mg | Verdinexor 40 mg
Number analyzed (Participants) | 5 | 6 | 6 | 6
Ratio | 0.9 | 1.0 | 1.1 | 1.1

14. Secondary Outcome: Accumulation Factor (AR) of AUC0-inf
Description: Accumulation factor was defined as a ratio of mean of AUC0-inf Day 3/ AUC0-inf Day 1 for plasma verdinexor.
Time Frame: Days 1 and 3: pre-dose, 15 minutes, 30 minutes, 1, 2, 3, 4, 8, 12, 24, 48 (only for Day 3) hours post-dose
Population: as for outcome 11
Measure: Number; unit: Ratio
Arm/Group | Verdinexor 5 mg | Verdinexor 10 mg | Verdinexor 20 mg | Verdinexor 40 mg
Number analyzed (Participants) | 5 | 6 | 6 | 6
Ratio | 0.9 | 1.0 | 1.1 | 1.0

15. Secondary Outcome: Maximum Tolerated Dose (MTD) of Verdinexor
Description: MTD was defined as the dose level tested in the cohort immediately preceding a cohort where one or more dose limiting toxicities (DLTs) were observed. A DLT was defined as any AE or abnormal laboratory value that the Investigator suspected was probably related to verdinexor that was severe in intensity or serious or Indicative of an unacceptable risk to additional participants in the study in the opinion of the Investigator or Sponsor.
Time Frame: From start of study drug administration up to Day 8
Population: MTD was not achieved at study completion due to early termination of study prior to observing protocol-specified DLT criteria. Therefore, no data was reported for this outcome measure.
Arm/Group | Placebo | Verdinexor 5 mg | Verdinexor 10 mg | Verdinexor 20 mg | Verdinexor 40 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to Day 33
Description: Safety population included all participants who received at least 1 dose of verdinexor or placebo.
Arm/Group | Placebo | Verdinexor 5 mg | Verdinexor 10 mg | Verdinexor 20 mg | Verdinexor 40 mg
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/8 | 6/6 | 3/6 | 4/6 | 5/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=8) | Verdinexor 5 mg (N=6) | Verdinexor 10 mg (N=6) | Verdinexor 20 mg (N=6) | Verdinexor 40 mg (N=6)
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 4
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Spermatozoa morphology abnormal (Investigations) | 0 | 0 | 0 | 1 | 1
Spermatozoa progressive motility decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 1 | 1 | 1
Dizziness postural (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 2 | 1 | 2 | 2
Lethargy (Nervous system disorders) | 0 | 3 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
This study was terminated due to administrative reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes